CLINICAL TRIAL: NCT01517035
Title: Peripheral Blood Stem Cell Allotransplantation for Hematological Malignancies Using Ex Vivo CD3, CD19 Depletion and CD34 Selection
Brief Title: Improving Blood Stem Cell Collection and Transplant Procedures
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 120028; 12-H-0028
Record Dates: First submitted 2012-01-24; First posted 2012-01-25 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2017-03-29

CONDITIONS: Myelodysplastic Syndrome (MDS); Chronic Myelogenous Leukemia; Acute Lymphoblastic Leukemia; CML (Chronic Myelogenous Leukemia; CLL (Chronic Lymphocytic Leukemia)
Keywords: Peripheral Blood Stem Cell Transplantation; Stem Cell Transplant; Transplant; Myelodyplastic Syndrome; MDS; Leukemia
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, B-Cell; Leukemia | interventions — Stem Cell Transplantation

ARMS (1):
- 1 (Experimental): Myeloablative conditioning (Flu/Cy/TBI) followed by CD3/19/34 selected stem cell graft.
  Interventions: Procedure: Stem Cell Transplantation

INTERVENTIONS:
Procedure: Stem Cell Transplantation — Myeloablative conditioning (Flu/Cy/TBI) followed by CD3/19/34 selected stem cell graft.

SUMMARY:
Background:

- People who have some kinds of cancer can benefit from donated bone marrow stem cells. These stem cells help produce healthy bone marrow and slow or stop the spread of abnormal cells. However, stem cells transplants do not always work. Also, they may have serious side effects that can cause illness or death. The Bone Marrow Stem Cell Transplant Program is studying methods to make stem cell transplant procedures safer and more effective.

Objectives:

- To test a new procedure that may improve the success and decrease the side effects of stem cell transplants.

Eligibility:

* Individuals 10 to 75 years of age who have a life-threatening illness that may require a stem cell transplant.
* Healthy siblings who are able to provide stem cells for transplant.

Design:

* Participants will be screened with a medical history, physical exam, and blood and urine tests.
* Donor procedures:
* Stem cell donors will start by having apheresis to donate white blood cells.
* Donors will receive filgrastim shots for 5 days to help move stem cells into the blood for collection.
* Donors will have another round of apheresis to donate the stem cells for transplant.
* Recipient procedures:
* Before the transplant, recipients will have radiation twice a day for 3 days and chemotherapy for 7 days.
* After the radiation and chemotherapy, recipients will receive the stem cells provided by the donor.
* After the transplant, recipients will receive the white blood cells provided by the donor.
* Recipients will be monitored closely for 4 months to study the success of the transplant. They will have more followup visits at least yearly thereafter.
* Recipients will have a research apheresis prior to transplant and at 3 months.

DETAILED DESCRIPTION:
Peripheral blood stem cell transplant research carried out by the NHLBI BMT Unit focus on transplant techniques designed to decrease graft versus host disease (GVHD), increase the graft-versus-leukemia (GVL) effect and reduce the risk of post-transplant graft rejection.

Through incremental transplant clinical trials we have shown that by controlling the stem cell (CD34+ cell) and T lymphocyte (CD3+ cell) dose, severe GVHD can be reduced whilst beneficial GVL effects can be preserved. We found that T cell depleted transplants using the Nexell/Baxter Isolex 300i system and subsequently, the Miltenyi CD34+ CliniMACs system to obtain high CD34+ doses depleted of lymphocytes were safe to administer and associated with less severe acute GVHD and promising response rates and overall survival. Our previous trials have helped us to create the transplant environment (significant lymphodepletion and minimal post transplant immunosuppression) that make for an ideal platform for adoptive cellular immunotherapy

This protocol is designed to evaluate the safety and efficacy of an improved ex vivo graft manipulation procedure using the Miltenyi CliniMACs CD 34, 3 and 19 selection system in HLA-matched sibling allogeneic peripheral blood stem cell transplant. The manipulation of the graft is the primary research intervention and all other aspects of clinical management on this protocol are the standard of care. The target CD34+ dose range will be 3 times 10(6)/kg to 10 times 10(6)/kg and the target CD3+ dose range will be 5 x 10(4)/kg to 1 times 10(6)/kg. The technique will preserve greater numbers of NK cells. Once we demonstrate adequacy of engraftment in the first ten recipients, we plan an amendment to permit further use of this protocol to serve as a platform for several planned adoptive cellular therapy initiatives.

The protocol will accrue up to 44 subjects aged 10-75 with a hematological malignancy and their HLA-matched sibling donors, in whom allogeneic stem cell transplantation from an HLA-matched sibling would be routinely indicated. Diagnostic categories will include acute and chronic leukemia, myelodysplastic syndromes, lymphomas, multiple myeloma and myeloproliferative syndromes.

Subjects will receive a myeloablative conditioning regimen of cyclophosphamide (120 mg/kg total), fludarabine (125 mg/m(2) total) and total body irradiation (1200 cGy with lung shielding to 600 cGy), followed by an infusion of a stem cell product prepared using the Miltenyi CliniMACS system for CD34, 3 & 19 selection. Older subjects will receive a lower dose of irradiation (600 cGy) without lung shielding to reduce the regimen intensity.

The overall objective is to assess the feasibility of using this system as a platform for cellular immunotherapy initiatives. The primary study endpoint will be overall survival at day plus 200. Non-relapse mortality at day plus 200 will be monitored for safety. Secondary endpoints will be standard transplant outcome variables such as non-hematologic toxicity, incidence and severity of acute and chronic GVHD and relapse of disease.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients in remission as well as patients with primary induction failure or refractory disease will be considered for inclusion. At the discretion of the PI, patients may continue standard of care treatment options to control their baseline disease burden up to the start of the protocol.

RECIPIENT

Ages 10-75 years inclusive

Chronic myelogenous leukemia (CML):

* Subjects under the age of 21 in chronic phase
* Subjects ages 10-75 in chronic phase who have failed treatment with imatinib, have intolerance to imatinib, or who did not receive imatinib at therapeutic doses within the first 12 months from diagnosis.
* Subjects ages 10-75 in accelerated phase or blast transformation.

Acute lymphoblastic leukemia (ALL): any of these categories: ALL in first remission with high-risk features (presenting leukocyte count >100,000/cu mm, Karyotypes t9; 22, t4, t19, t11, biphenotypic leukemia) All second or subsequent remissions, primary induction failure, partially responding or untreated relapse.

Acute myelogenous leukemia (AML): AML in first remission - except AML with good risk karyotypes: AML M3 (t15; 17), AML M4Eo (inv 16), AML t (8; 21). All AML in second or subsequent remission, primary induction failure and resistant relapse.

Myelodysplastic syndromes(MDS): any of these categories - refractory anemia with transfusion dependence, refractory anemia with excess of blasts, transformation to acute leukemia, chronic myelomonocytic leukemia, atypical MDS/myeloproliferative syndromes.

Myeloproliferative disorders including atypical (Ph negative) chronic myeloid and neutrophilic leukemias, progressing myelofibrosis, and polycythemia vera, essential thrombocythemia in transformation to acute leukemia or with progressive transfusion requirements or pancytopenia.

Chronic lymphocytic leukemia refractory to fludarabine treatment and with bulky progressive disease or with thrombocytopenia (less than or equal to 100,000/ micro-l) or anemia (less than or equal to 10g/dl) not due to recent chemotherapy.

Non-Hodgkin s lymphoma including Mantle cell lymphoma relapsing or refractory to standard of care treatments.

Multiple myeloma, Waldenstroms macroglobulinemia, unresponsive or relapsed following standard of care treatments.

HLA identical (6/6) related donor.

For adults: Ability to comprehend the investigational nature of the study and provide informed consent. For minors: written informed consent from one parent or guardian. Informed oral consent from minors: the process will be explained to the minor on a level of complexity appropriate for their age and ability to comprehend.

DONOR

Related donor, HLA identical (6/6) with recipient

Weight greater than or equal to 18 kg

Age greater than or equal to 2 or less than or equal to 80 years old

For adults: Ability to comprehend the investigational nature of the study and provide informed consent. For minors: Written informed consent from one parent or guardian and informed assent: The process will be explained to the minor on a level of complexity appropriate for their age and ability to comprehend.

EXCLUSION CRITERIA:

RECIPIENT (any of the following)

Estimated probability of surviving less than three months

Major anticipated illness or organ failure incompatible with survival from transplant

Severe psychiatric illness. Mental deficiency sufficiently severe as to make compliance with the transplant treatment unlikely and making informed consent impossible.

Positive pregnancy test for women of childbearing age.

HIV positive

DLCO adjusted for Hb and ventilation < 50% predicted

Left ventricular ejection fraction < 40% (evaluated by ECHO) or < 30% (evaluated by MUGA)

AST/SGOT > 10 times ULN (>grade 3, CTCAE)

Bilirubin > 5 times ULN (>grade 3, CTCAE)

Creatinine > 4.5 times ULN (>grade 3, CTCAE)

Prior allogeneic stem cell transplantation

DONOR (any of the following)

Pregnant or breast-feeding. Lactating donors are permitted provided breastmilk is discarded during the days filgatrim (G-CSF) is given.

Unfit to receive G-CSF and undergo apheresis (abnormal blood counts, history of stroke, uncontrolled hypertension)

Sickling hemaglobinopathy including HbSS, HbAS, HbSC

Donors who are positive for HIV active hepatitis B (HBV), hepatitis C (HCV) or human T-cell lymphotropic virus (HTLV-I/II)

Severe psychiatric illness. Mental deficiency sufficiently severe as to make compliance with the BMT treatment unlikely, and making informed consent impossible.

Age greater than or equal to 80 years old

Children who weigh less than or equal to 18 kg and are < 2 years of age.

Ages: 2 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2012-01-13; Primary Completion 2017-03-29 (Actual); Study Completion 2017-03-29 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is all cause mortality at day 200, and the proportion of subjects who have survived at day 200 will be used to determine the sample size. | 200 days

SECONDARY OUTCOMES:
Cumulative incidence of relapse | 3 years
Secondary Outcome Measure: Standard transplant outcome variables such as relapse, non-relapse mortality, neutrophil and platelet recovery kinetics, incidence and severity of acute GVHD and chronic GVHD. Technical success rates and the use of DLI...
Non Relapse Mortality | 3 years
Days till ANC greater than 500/uL | variable
Days till Platelet greater than 20 k/ul | variable

CONTACTS AND LOCATIONS:
Overall Officials: Minocher M Battiwalla, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Muller AM, Linderman JA, Florek M, Miklos D, Shizuru JA. Allogeneic T cells impair engraftment and hematopoiesis after stem cell transplantation. Proc Natl Acad Sci U S A. 2010 Aug 17;107(33):14721-6. doi: 10.1073/pnas.1009220107. Epub 2010 Aug 2. PMID 20679222
- [Background] Maury S, Lemoine FM, Hicheri Y, Rosenzwajg M, Badoual C, Cherai M, Beaumont JL, Azar N, Dhedin N, Sirvent A, Buzyn A, Rubio MT, Vigouroux S, Montagne O, Bories D, Roudot-Thoraval F, Vernant JP, Cordonnier C, Klatzmann D, Cohen JL. CD4+CD25+ regulatory T cell depletion improves the graft-versus-tumor effect of donor lymphocytes after allogeneic hematopoietic stem cell transplantation. Sci Transl Med. 2010 Jul 21;2(41):41ra52. doi: 10.1126/scitranslmed.3001302. PMID 20650872
- [Background] Thomson KJ, Morris EC, Milligan D, Parker AN, Hunter AE, Cook G, Bloor AJ, Clark F, Kazmi M, Linch DC, Chakraverty R, Peggs KS, Mackinnon S. T-cell-depleted reduced-intensity transplantation followed by donor leukocyte infusions to promote graft-versus-lymphoma activity results in excellent long-term survival in patients with multiply relapsed follicular lymphoma. J Clin Oncol. 2010 Aug 10;28(23):3695-700. doi: 10.1200/JCO.2009.26.9100. Epub 2010 Jul 6. PMID 20606089